CLINICAL TRIAL: NCT01061684
Title: Nonalcoholic Fatty Liver Disease (NAFLD) Pediatric Database 2
Brief Title: NAFLD Pediatric Database 2
Acronym: NAFLD Peds DB2
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: NAFLD Pediatric Database 2; U01DK061730 (NIH)
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Liver Disease
Keywords: fatty liver disease; NASH; NAFLD; non-alcoholic steatohepatitis
MeSH Terms: conditions — Liver Diseases; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, liver tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NAFLD: pediatric patients with non-alcoholic fatty liver disease (NAFLD).

SUMMARY:
The NAFLD Database 2 will recruit at least 650 new pediatric participants with liver biopsies and contemporaneous biosamples, and will also invite pediatric participants from the prior NAFLD Database and TONIC trial (50 with a recent biopsy and 150 without a contemporaneous biopsy) to enroll in the NAFLD Pediatric Database 2 study. Combining the new and continuing participants leads to a recruitment goal for the pediatric Database 2 of 850 pediatric participants during the enrollment period.

DETAILED DESCRIPTION:
All the new pediatric participants will have had a liver biopsy within 120 days prior to enrollment coupled with contemporaneous biosamples within 90 days prior to enrollment and up to 90 days before or 4-90 days after the biopsy. We estimate that at least 50 of the continuing pediatric participants will be due for a standard of care liver biopsy at the time of their enrollment into the pediatric Database 2 study, and will, as a result, also have a liver biopsy and contemporaneous biosamples.

ELIGIBILITY:
Inclusion Criteria:

* Continuing participants:

  * Previously enrolled in the NAFLD Database study or TONIC trial
  * Age at least 2 years and not older than 17 years during the consent process
  * Willingness to continue to be followed for up to 4 years
  * Ability and willingness to give written, informed parental consent and child assent, per local IRB guidelines, to be enrolled into the pediatric Database 2 study
* New participants:

  * Age at least 2 years of age and not older than 17 years during the consent process
  * Willingness to be followed for up to 4 years
  * Ability and willingness to give written, informed parent consent and child assent to be enrolled into the pediatric Database 2 study
  * Minimal or no alcohol use history consistent with NAFLD
  * Having undergone a liver biopsy that is obtained within 120 days of enrollment
  * Collection of biosamples (serum, plasma, DNA, and, if available, liver tissue) within 90 days prior to enrollment and 0-90 days before or 4-90 days after the standard of care liver biopsy

Exclusion Criteria:

* Total parenteral nutrition for more than 1 month within a 6 month period before baseline liver biopsy
* Short bowel syndrome
* History of gastric or jejunoileal bypass preceding the diagnosis of NAFLD. Bariatric surgery performed following enrollment is not exclusionary. Liver biopsies obtained during bariatric surgery cannot be used for enrollment because of the associated surgical or anesthetic acute changes and the weight loss efforts that precede bariatric surgery
* History of biliopancreatic diversion
* Evidence of advanced liver disease defined as a Child-Pugh-Turcotte score equal to or greater than 10
* Evidence of chronic hepatitis B as marked by the presence of HBsAg in serum (participants with isolated antibody to hepatitis B core antigen, anti-HBc total, are not excluded)
* Evidence of chronic hepatitis C as marked by the presence of anti-HCV or HCV RNA in serum
* Low alpha-1-antitrypsin level and ZZ phenotype (both determined at the discretion of the investigator)
* Wilson's disease
* Known glycogen storage disease
* Known dysbetalipoproteinemia
* Known phenotypic hemochromatosis (HII greater than 1.9 or removal of more than 4 g of iron by phlebotomy)
* Prominent bile duct injury (florid duct lesions or periductal sclerosis) or bile duct paucity
* Chronic cholestasis
* Vascular lesions (vasculitis, cardiac sclerosis, acute or chronic Budd-Chiari, hepatoportal sclerosis, peliosis)
* Iron overload greater than 3+
* Zones of confluent necrosis, infarction, massive or sub-massive, pan-acinar necrosis
* Multiple epithelioid granulomas
* Congenital hepatic fibrosis
* Cystic fibrosis
* Polycystic liver disease
* Other metabolic or congenital liver disease
* Evidence of systemic infectious disease
* Known HIV positive
* Disseminated or advanced malignancy
* Concomitant severe underlying systemic illness that in the opinion of the investigator would interfere with completion of follow-up
* Active drug use or dependence that, in the opinion of the study investigator, would interfere with adherence to study requirements
* Any other condition, which in the opinion of the investigator would impede compliance or hinder completion of study
* Inability for parent to provide informed consent and child 8 years or greater to give assent

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants at least 2 years of age and less than 18 years of age with known or suspected NAFLD or NASH-related cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 969 (Actual)
Dates: Start 2010-01-20 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Liver histology scores | varies
  Liver histology scores (derived from central reading of liver biopsy at entry, standard of care biopsy done during screening or follow-up, or liver biopsy obtained for the TONIC trial)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (12):
- United States (12):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago (NWU), Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - St. Louis University, St Louis, Missouri
  - University at Buffalo-Women and Children's Hospital of Buffalo, Buffalo, New York
  - Columbia University, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital- UW, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to www.niddkrepository.org at the end of the funding.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available once the funding cycle ends.
Access Criteria: Access requires registration and approval from the NIDDK Repository.
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- [Derived] Rausch JC, Lavine JE, Chalasani N, Guo X, Kwon S, Schwimmer JB, Molleston JP, Loomba R, Brunt EM, Chen YI, Goodarzi MO, Taylor KD, Yates KP, Rotter JI; NASH Clinical Research Network. Genetic Variants Associated With Obesity and Insulin Resistance in Hispanic Boys With Nonalcoholic Fatty Liver Disease. J Pediatr Gastroenterol Nutr. 2018 May;66(5):789-796. doi: 10.1097/MPG.0000000000001926. PMID 29470286
- [Derived] Molleston JP, Schwimmer JB, Yates KP, Murray KF, Cummings OW, Lavine JE, Brunt EM, Scheimann AO, Unalp-Arida A; NASH Clinical Research Network. Histological abnormalities in children with nonalcoholic fatty liver disease and normal or mildly elevated alanine aminotransferase levels. J Pediatr. 2014 Apr;164(4):707-713.e3. doi: 10.1016/j.jpeds.2013.10.071. Epub 2013 Dec 19. PMID 24360992
- See also: Nonalcoholic Steatohepatitis Clinical Research Consortium — https://jhuccs1.us/nash/
- See also: The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) — http://www2.niddk.nih.gov/